CLINICAL TRIAL: NCT01709734
Title: ARMOR2: A 2 Part, Phase 2 Trial of Galeterone in the Treatment of Castration Resistant Prostate Cancer
Brief Title: A 2 Part, Phase 2 Trial of Galeterone in the Treatment of Castration Resistant Prostate Cancer
Acronym: ARMOR2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated prematurely in all investigational study centers upon recommendation from the study's Data Monitoring Committee (DMC).
  Study was stopped due to lack of efficacy.
Sponsor: LTN PHARMACEUTICALS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOK-200-10
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-hydroxy-17-(1H-benzimidazole-1-yl)androsta-5,16-diene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Confirmation (Experimental): Dose A - galeterone tablets once daily PO for three months + extension
  Dose B - galeterone tablets once daily PO for three months + extension
  Dose C - galeterone tablets once daily PO for three months + extension
  Interventions: Drug: galeterone
- Dose Expansion (Experimental): Single dose expansion (from part 1) of galeterone tablets once daily PO for three months + extension
  Interventions: Drug: galeterone

INTERVENTIONS:
Drug: galeterone
  Other Names: TOK-001

SUMMARY:
A Phase 2, 2 part trial to evaluate the safety and efficacy of galeterone in castration resistant prostate cancer (CRPC) patients.

DETAILED DESCRIPTION:
This trial will be split into two parts. The purpose of Part 1 will be to confirm dose and target patient population and Part 2 will be expansion of the dose and patient population selected in Part 1. For eligible patients, there will be an optional extension dosing following the completion of Part 1 or Part 2 of the trial.

Obtaining of informed consent and screening may be performed up to 28 days prior to enrollment. Each patient will be able to receive his specified regimen for 3 consecutive cycles. Each cycle consists of 28 days (approximately 1 mo.). End of Cycle 3 visit assessments will be used to determine outcome and dosing may continue up to an additional 2 weeks until the results of all assessments are obtained. Eligible patients may continue treatment in an optional extension period following the completion of the primary parts of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate
2. Ongoing androgen blockade demonstrated by serum testosterone concentration of less than 50 ng/dL
3. Demonstration of progression while on androgen blockade
4. Eastern Cooperative Oncology Group (ECOG) Performance Status <2

Exclusion Criteria:

1. Depending upon patient prior treatment the following apply:

   * Prior treatment with CYP17 inhibitors or AR antagonists (e.g. abiraterone, TAK-700, ARN-509, ketoconazole*, enzalutamide, or galeterone) - Treatment naïve only
   * Prior treatment with CYP17 inhibitors (e.g. TAK-700, ketoconazole*) or AR antagonists (e.g. enzalutamide, ARN-509,) or galeterone - abiraterone refractory only
   * Prior treatment with CYP17 inhibitors (e.g. abiraterone, TAK-700, ketoconazole*) or AR antagonists (e.g. ARN -509) or galeterone - enzalutamide refractory only
2. Prior chemotherapy (unless allowed for some study arms)
3. Treatment with non-steroidal oral antiandrogens within 4 weeks of enrollment
4. Prior use of any chronic systemic glucocorticoids .
5. Prior radiation therapy within 3 weeks and radionuclide therapy within 8 weeks of enrollment
6. Prior treatment with Alpharadin® (Xofigo®)
7. Treatment with anti arrhythmia therapy for ventricular arrhythmia < 4 weeks prior to enrollment
8. Treatment with Coumadin® or other anti-coagulant therapy (except aspirin) < 4 weeks prior to enrollment
9. Severe systemic diseases or active uncontrolled illnesses.
10. Abnormal heart function
11. Liver metastases
12. Brain metastases (unless stable disease >3 mos. by scan without additional CNS-directed therapy)
13. The patient has known allergy to any of the treatment components
14. Any physical or mental condition or social situation that in the opinion of the Investigator may interfere with the patient's ability to comply with the trial procedures
15. History of excessive alcohol consumption
16. Use of any substance known to cause AME

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Confirmation of recommended dose and patient population for Part 2 of the study. | 3 months
  Confirmation of recommended dose and patient population for Part 2 of the study.
Assessment of efficacy by means of PSA response. | 3 months
  Assessment of efficacy by means of PSA response.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, M.D., Principal Investigator — University of Washington Seattle Cancer Care Alliance; Mary Ellen Taplin, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (23):
- United States (21):
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Tulane Cancer Center, New Orleans, Louisiana
  - AAHS Research Institute, Annapolis, Maryland
  - University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Coastal Urology Associates, Brick, New Jersey
  - Premier Urology Associates, LLC, Lawrenceville, New Jersey
  - Roswell Park Center Institute, Buffalo, New York
  - Mount Sinai, New York, New York
  - Carolina Clinical Trials, Concord, North Carolina
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario